CLINICAL TRIAL: NCT01278121
Title: Food and Health; Testing of the Anti-Inflammatory Potential of a Macronutrient Balanced Normocaloric Diet
Brief Title: Study of the Potential of a Macronutrient Balanced Normocaloric Diet to Treat Lifestyle Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010.1122.3
Record Dates: First submitted 2010-07-04; First posted 2011-01-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Obesity; Diabetes Mellitus, Type 2; Cardiovascular diseases
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Adiposity; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet A: High-fat diet (Other): Diet given for 3 days to "reset" all of the participants
  Interventions: Dietary Supplement: Diet A
- Diet B: A carbohydrate-restricted diet (Active Comparator): The diet will be given for 10 days, 6 meals a day
  Interventions: Dietary Supplement: Diet B

INTERVENTIONS:
Dietary Supplement: Diet A — 3 days, 6 meals a day
  Other Names: Diet intervention; Obesity
  Arms: Diet A: High-fat diet
Dietary Supplement: Diet B — 10 days, 6 meals a day
  Other Names: Low carbohydrate diet
  Arms: Diet B: A carbohydrate-restricted diet

SUMMARY:
One of today's major health problem in the western world is related to lifestyle. Lifestyle diseases include obesity, type 2 diabetes, cardiovascular diseases and different types of cancers. For many years, a low-fat diet has been recommended to reduce obesity and lifestyle diseases, but replacing fat with carbohydrates has lead to an increase of these diseases. Overweight is associated with a chronical low-degree inflammation, and later studies have shown that carbohydrates have an effect on the mechanisms of inflammation. Previous studies in the investigators group has shown that in healthy, but slightly overweight persons, a balanced diet of lower carbohydrate content regulates the gene expression in a manner that leads to less inflammation. In this study the investigators will look at morbid obese women (BMI>35) to see if the same, balanced diet can improve the inflammatory profile of the women.

DETAILED DESCRIPTION:
The hypothesis of this proposal is that a carbohydrate-rich diet may cause a major deregulation of hormonal balance, causing both acute and chronic systemic inflammatory reactions mediated by white blood cells. We furthermore postulate that a carbohydrate-rich diet is a major risk factor in the development of obesity and life style diseases directly resulting from chronic systemic inflammation. We therefore want to use an integrated multidisciplinary systems biology approach to identify the hormones, genes and pathways specifically responding to a dietary carbohydrate reduction, to develop biomarkers that can be used for risk assessment, to identify molecular pathways and build mathematical models that describe the link between diet and inflammation, and use this knowledge to provide personalised dietary advice.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 kg/m2

Exclusion Criteria:

* Allergies (fish, nuts, eggs)
* Patient under treatment/using medicine that can influence results
* Pregnancy and lactation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in microarray gene expression | Day 1, 4 and 14
  Changes in microarray gene expression profiles in blood from morbid obese women, in response to balanced dietary macro nutrient composition

SECONDARY OUTCOMES:
Inflammatory markers, hormonal dietary responses and blood lipids | Day 1, 4 and 14
  Blood will be screened for hormones, blood lipids and other inflammatory biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Berit Johansen, PhD, Principal Investigator — Norwegian University of Science and Technology; Marian Forde, Cand.Scient., Study Chair — Norwegian University of Science and Technology
Locations (1):
- NTNU Department of Biology, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Brattbakk HR, Arbo I, Aagaard S, Lindseth I, de Soysa AK, Langaas M, Kulseng B, Lindberg F, Johansen B. Balanced caloric macronutrient composition downregulates immunological gene expression in human blood cells-adipose tissue diverges. OMICS. 2013 Jan;17(1):41-52. doi: 10.1089/omi.2010.0124. Epub 2011 Jun 16. PMID 21679058